CLINICAL TRIAL: NCT00339560
Title: A Population-Based Case-Control Study of Biliary Tract Cancers in Shanghai, China
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999997028; OH97-C-N028
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Biliary Tract Cancer
Keywords: Ampulla of Vater; Gallbaldder; Cancer; Extrahepatic Bile Duct
MeSH Terms: conditions — Biliary Tract Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Cases will bile duct CA: Patients with bile duct cancer
- Cases with Gallbladder CA: Patients with gallbladder cancer
- Controls with gall stones: Patients undergoing cholecystectomy for gall stones
- Controls without cancer: Hospital controls with cancer

SUMMARY:
The key aims of this study include estimation of possible risk associated with a history of gallstones, bacterial infection for the biliary tract, other medical history, diet, use of tobacco and alcohol, obesity, reproductive factors, and family history of cancer. Information will be used to examine risk patterns a) seperately by anatomic subsite; b) among patients with gallbladder cancer vs. controls undergoing cholecystectomy for gallstones; c) among the patients with bile duct cancer vs. Hospital controls without cancer who undergo surgery for removal of bile duct stones. We will also attempt to ascertain reasons for cancer who undergo surgery for removal of bile duct stones. We will also attempt to ascertain reasons for the rising incidence of biliary tract cancers in Shanghai. Serum collected from all subjects will be analyzed for estrogens and other hormones, vitamins C and E, cholesterol, and bacterial antibodies (including salmonella typhi, paratyphi, and escherischia coli). Bile fluid will be cultured for aerobic bacteria, and gallstones analyzed for color, cholesterol, and evidence of bacteria infection. A major challenge in biliary tract cancer research is to determine how cancer risk factors differ from those for gallstones or biliary duct stone disease, since many people have gallstones (or biliary duct stones) but few develop cancer....

DETAILED DESCRIPTION:
The key aims of this study include estimation of possible risk associated with a history of gallstones, bacterial infection for the biliary tract, other medical history, diet, use of tobacco and alcohol, obesity, reproductive factors, and family history of cancer. Information will be used to examine risk patterns a) seperately by anatomic subsite; b) among patients with gallbladder cancer vs. controls undergoing cholecystectomy for gallstones; c) among the patients with bile duct cancer vs. Hospital controls without cancer who undergo surgery for removal of bile duct stones. We will also attempt to ascertain reasons for cancer who undergo surgery for removal of bile duct stones. We will also attempt to ascertain reasons for the rising incidence of biliary tract cancers in Shanghai. Serum collected from all subjects will be analyzed for estrogens and other hormones, vitamins C and E, cholesterol, and bacterial antibodies (including salmonella typhi, paratyphi, and escherischia coli). Bile fluid will be cultured for aerobic bacteria, and gallstones analyzed for color, cholesterol, and evidence of bacteria infection. A major challenge in biliary tract cancer research is to determine how cancer risk factors differ from those for gallstones or biliary duct stone disease, since many people have gallstones (or biliary duct stones) but few develop cancer.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cases of biliary tract cancer newly diagnosed between September 1, 1996 and August 31, 1999 among residents of urban Shanghai.

Must be under the age of 75 at the time of diagnosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of Shanghai.
Sampling Method: Non-Probability Sample
Enrollment: 2624 (Actual)
Dates: Start 1997-05-16 (Actual); Primary Completion 2008-05-21 (Actual); Study Completion 2008-05-21 (Actual)

PRIMARY OUTCOMES:
Gallbladder Cancer | 5 years
  Gallbladder cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jill E. Koshiol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Shanghai Cancer Institute, Shanghai, China

REFERENCES:
- [Background] Strom BL, Hibberd PL, Soper KA, Stolley PD, Nelson WL. International variations in epidemiology of cancers of the extrahepatic biliary tract. Cancer Res. 1985 Oct;45(10):5165-8. PMID 4027991
- [Background] Jin F, Devesa SS, Zheng W, Blot WJ, Fraumeni JF Jr, Gao YT. Cancer incidence trends in urban Shanghai, 1972-1989. Int J Cancer. 1993 Mar 12;53(5):764-70. doi: 10.1002/ijc.2910530510. PMID 8449600
- [Background] Devesa SS, Silverman DT, Young JL Jr, Pollack ES, Brown CC, Horm JW, Percy CL, Myers MH, McKay FW, Fraumeni JF Jr. Cancer incidence and mortality trends among whites in the United States, 1947-84. J Natl Cancer Inst. 1987 Oct;79(4):701-70. PMID 3309421